CLINICAL TRIAL: NCT03857672
Title: The Efficacy of Hypnotic Cognitive Therapy for Chronic Pain in SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Charles Bombardier, Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004135; 534402 (Other: Craig H. Neilsen Foundation)
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries; Chronic Pain
Keywords: Behavioral; Cognitive Therapy; Self-Hypnosis
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators will conceal treatment group assignment from staff that conduct outcome assessments by: using a permuted blocked randomization with random block sizes, using secure email to inform the interventionist about group assignment, keeping the interventionist and outcome assessor physically separate and sound isolated in research spaces, and training staff in other day-to-day measures designed to maintain the blind. Research staff will be educated about the importance of maintaining the blinded conditions of the study and strategies to engage participants in maintaining the blinding as well (being clear about who participants contact regarding study questions, reminding participants about maintaining the secrecy of their condition at the beginning of all outcome related calls, having the therapist remind participants to keep their condition secret from staff assessing outcomes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotic Cognitive Therapy (HYPNOCT) (Experimental): The HYPNOCT arm will use hypnotic strategies and suggestions for identifying adaptive cognitions and for making adaptive changes in cognitions more integrated into the participant's belief system (note that traditional CT uses purposeful argument and logic to make these changes; in this condition the investigators add a hypnotic automaticity to this process). Thus, HYPNOCT is a hybrid intervention that overlaps with both hypnosis and CT. The participant will relax in a comfortable position and listen to the clinician speak. However, unlike standard hypnosis for pain, the post-induction suggestions will focus on changes in cognitive content and processes (as opposed to changes in sensory experience). The participants will undergo 6 weekly sessions each lasting 30-40 minutes.
  Interventions: Behavioral: Hypnotic Cognitive Therapy (HYPNOCT)
- Usual Care (No Intervention): The study therapist will notify participants assigned to Usual Care via the participant's preferred mode of communication (phone, U.S. mail, or email). People assigned to usual care will be encouraged to continue using the health care services available to them to address their pain. The study therapist will emphasize the importance of completing the outcome assessments. The treatments usual care participants actually received will be assessed at 6 and 12 weeks.

INTERVENTIONS:
Behavioral: Hypnotic Cognitive Therapy (HYPNOCT) — The HYPNOCT intervention will use hypnotic strategies and suggestions for identifying adaptive cognitions and for making adaptive changes in cognitions more integrated into the participant's belief system (note that traditional CT uses purposeful argument and logic to make these changes; in this condition the investigators add a hypnotic automaticity to this process). Thus, HYPNOCT is a hybrid intervention (more than the sum of CT and hypnosis) that overlaps with both hypnosis and CT. The participant will relax in a comfortable position and listen to the clinician speak. However, unlike standard hypnosis for pain, the post-induction suggestions will focus on changes in cognitive content and processes (as opposed to changes in sensory experience).
  Arms: Hypnotic Cognitive Therapy (HYPNOCT)

SUMMARY:
Chronic pain is prevalent and disabling in people with spinal cord injury (SCI). Medications alone often do not cure the pain. Pilot research suggests that training in the combination of self-hypnosis and cognitive therapy (HCT) can reduce chronic SCI-related pain. Thus far, people have learned HCT only through in-person training sessions plus home practice. The investigators think that training in HCT could be as effective if the training is done via videoconferencing. The purpose of this study is to find out whether people who are trained in HCT via videoconferencing achieve significant pain relief and other benefits compared to people who receive usual medical care (UC) for pain. Bettering our understanding of videoconferencing-delivered HYPNOCT can greatly increase treatment accessibility for individuals with SCI.

Aim 1: To compare the efficacy of HYPNOCT vs. UC in adults with SCI and chronic pain. Investigators will compare the effect of the intervention on patient-reported average daily pain as measured by a 0-10 numerical rating scale.

Aim 2: To examine sex, race/ethnicity, and pain type (neuropathic vs. non-neuropathic) as potential effect modifiers.

Hypotheses Primary study hypothesis Hypothesis 1a: There will be a significantly greater reduction in average daily pain intensity from baseline to the end of treatment in the HYPNOCT group compared to the UC group.

Secondary study hypotheses Hypothesis 1b: Compared to the UC group, participants in the HYPNOCT group will show greater improvement in pain interference, depression, sleep quality, subjective disability, health-related quality of life, community participation, pain catastrophizing, pain acceptance, and global improvement.

Hypothesis 2: The investigators will examine whether sex, race/ethnicity, and pain type (neuropathic vs. non-neuropathic) exert a modifying effect upon outcomes.

DETAILED DESCRIPTION:
This is a two-group randomized controlled trial designed to determine whether videoconferencing-delivered, hypnosis enhanced cognitive therapy (HYPNOCT) is an effective treatment for chronic SCI-related pain compared to usual care (UC). Those who consent to participate in the study will be randomized to HYPNOCT or UC. Following enrollment, but prior to starting treatment, participants will be assessed via three short (1 minute) interviews and one long (30-40 minutes) interview within a period of seven days. The assessments will also be administered immediately following the end of treatment (Post-treatment, after weekly session #6) and 6 weeks following the end of treatment (12 week follow-up) for a total of three assessment time points. The post-treatment assessments will also include additional questions related to treatment. The study has two aims.

Primary Objective: This trial is designed to assess whether videoconferencing-delivered, hypnosis enhanced cognitive therapy (HYPNOCT) is an effective treatment for chronic SCI-related pain compared to usual care (UC). Efficacy will be determined by comparing average pain intensity between the two groups at the end of the 6-week treatment phase, after controlling for baseline pain intensity and any confounders.

Hypothesis 1a: There will be a significantly greater reduction in average daily pain intensity from baseline to the end of treatment (6 weeks) in the HYPNOCT group compared to the UC group.

Secondary analyses will examine whether HYPNOCT and UC differ on pain interference, depression, sleep quality, subjective disability, health-related quality of life, and community participation at the end of treatment as well as at 12-week follow-up. Pain medications will be assessed at all time points and may be included as a covariate in outcome analyses.

Hypothesis 1b: Compared to the UC condition, the HYPNOCT condition will demonstrate significantly greater improvement on secondary outcomes (pain interference, depression, sleep quality, subjective disability, health-related quality of life, community participation, pain catastrophizing, pain acceptance, and global improvement) at 6 weeks and on the primary and secondary outcomes at 12 weeks.

Hypothesis 2: This is an exploratory hypothesis. The investigators will examine whether sex, race/ethnicity, and pain type (neuropathic vs. non-neuropathic) are effect modifiers.

Design and Outcomes A single center, randomized, single blind 160 subject efficacy study comparing videconferencing-delivered hypnosis-enhanced cognitive therapy (HCT) and usual care (UC) for the treatment of chronic SCI pain.

Interventions and Duration Participants will undergo a baseline assessment and then be randomized 1:1 to 6 weekly sessions of HYPNOCT vs. UC. Those in the HYPNOCT condition will have a weekly video-conference session with the study therapist over the course of 6 weeks. Each session will last between 45 and 60 minutes. Those in the UC condition will continue their usual care and receive no additional training from the study. The primary outcome assessment will be conducted at 6 weeks post-randomization. A follow-up assessment will be conducted in a similar manner at 12 weeks post-randomization. The primary outcome will be average pain intensity rated on a 1-10 numerical analog scale assessed four times within a one-week period.

For participants, the duration of the study will be approximately 3 to 4 months.

Sample Size and Population Researchers plan to enroll 160 participants with moderate to severe SCI-related chronic pain. Enrolled patients who complete the baseline assessments will be randomized into the HYPNOCT or UC conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older;
2. diagnosis of SCI at any level or severity;
3. completed inpatient rehabilitation (to ensure diagnosis and sufficient severity of SCI);
4. of ≥ 4 on a 0-10 NRS of pain intensity in the last week (during both the screening and baseline examinations)
5. reports that pain interferes with general activities (rates pain interference ≥ 1 on 0-10 scale)
6. reports pain has been present 12 weeks or more (chronic);
7. reports being able to read and speak English.
8. Have access to a webcam & microphone through either a computer, smartphone, or other internet-connected device.

Exclusion Criteria:

1. Severe cognitive impairment defined as one or more errors on the Six-Item Screener;
2. presence or history of mental health problems that would require referral for more intensive treatment or complicate hypnotic treatment (current suicidal ideation with intent or plan to harm oneself, current drug or alcohol dependence, lifetime history of bipolar disorder, psychosis, paranoid disorder based on screening questions from the M.I.N.I Neuropsychiatric Interview;
3. primary chronic pain problem pre-dated SCI (e.g., chronic headache);
4. has not undergone a previous medical evaluation for their pain to rule out treatable causes or undiagnosed disease (e.g., cancer);
5. unstable pain medication regimen (dosage changes within the past 3 weeks);
6. currently receiving CT or hypnosis for pain or has failed prior treatment with CT or hypnosis; and
7. declines to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Average Pain Intensity | Assessed via telepone four times within a 1-week period at baseline (prior to randomization), and at 6 and 12 weeks following randomization.
  Change in average pain intensity will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their pain intensity. Higher scores indicate higher levels of self-reported pain intensity.

SECONDARY OUTCOMES:
Change in Pain interference | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in pain interference will be measured using the Brief Pain Interference Scale which examines pain interference in 7 life domains within the past week. Responses for each item will be summed for a total raw score from 0 to 70. Higher scores indicate more self-reported pain interference.
Change in Depression | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in number and frequency of depressive symptoms will be measured with the Patient Health Questionnaire-9 (PHQ-9). Responses for each item will be summed for a total raw score from 0 to 27. Higher scores indicate more self-reported levels of depressive symptoms.
Change in Subjective Disability | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in subjective disability will be measured with the Sheehan Disability Scale to determine how SCI disrupts work/school, social life or family life/home responsibilities. Responses for each item will be summed for a total score from 0 to 30. Higher scores indicate more self-reported levels of subjective disability.
Change in Satisfaction with Life | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  The inves will use the 10-item SCIQOL Satisfaction with Social Roles and Activities-Short Form to measure this domain because this measure was recently developed specifically for persons with SCI. Five items are reversed coded. All responses from items are summed into a total score. Higher scores indicate higher self-reported satisfaction with life.
Change in Community Participation | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  The investigators will use the SCIQOL Ability to Participate short form to measure community participation because this measure was recently developed specifically for persons with SCI. Responses from items will be summed into a total score. Higher scores indicate higher levels of self-reported community participation.
Change in Pain Catastrophizing | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in pain catastrophizing will be measured with the 13-item Sullivan's Pain Catastrophizing Scale. Responses from each item will be summed for a total score from 0 to 52. Higher scores indicate higher levels of self-reported pain catastrophizing.
Change in Pain Acceptance | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in pain acceptance (positive coping concept) will be measured with the 8-item Chronic Pain Acceptance Questionnaire. Items 4, 5, 7, and 8 are reverse scored. All item responses are summed for a total score, with higher scores denoting higher levels of self-reported pain acceptance.
Change in Sleep Quality | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in sleep quality will be measured with the PROMIS-Sleep Disturbance Short Form 8a. The item responses are them summed and multiplied by the total number of items in the short form. Then this is divided by the number of items that were answered to get a prorated raw score. The pro-rated score is converted into a T-score for each participant which rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more self-reported sleep disturbance.
Change in Pain Self Efficacy | Assessed via telephone interview at baseline prior to randomization, and at 6 and 12 weeks following randomization.
  Change in pain self-efficacy will be assessed using the 4-item Patient Self-Efficacy Questionnaire (PSEQ). Responses from each item will be summed for a total score. Greater scores represent higher self-reported pain self-efficacy.
Change in Global Improvement Treatment Satisfaction | Assessed via telephone interview at 6 and 12 weeks following randomization.
  Assessed using the Patient Global Impression of Importance of Change and the Patient Global Assessment of Treatment Satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bombardier, PhD, Principal Investigator — University of Washington
Locations (1):
- Rehabilitation Medicine, Harborview Medical Center, Seattle, Washington, United States